## Effect of in vitro fertilisation (IVF) hormonal therapy on metabolic, endocrine and inflammatory status in IVF-conceived pregnancy

NCT03426228

## **Informed Consent Form**

Project: Effect of in vitro fertilisation (IVF) hormonal therapy on metabolic, endocrine and inflammatory status in IVF-conceived pregnancy

وغيرها من الانسولين ومقاومة الجلوكوز على توازن الإخصاب أدوية تأثير :دراسة مشروع المؤشرات الأيضية لدى المرضى الذين يخضعون لعلاج أطفال الانابيب

The United Arab Emirates (U.A.E) are listed among the top 10 countries worldwide in term of obesity and have one of the highest rates of polycystic ovary syndrome (PCOS), whereby 60% of Gulf women and 30% of Indian origins women living in the U.A.E have PCOS. Obesity has increased along with increasing related abnormalities in the reproductive system, such as an ovulation and infertility. In fact, 20% of couples worldwide are infertile; this corresponds to 50% of women in the UAE are facing infertility issues. Obesity is considered as a major risk factor for developing pregnancy-related complications such as gestational diabetes (GDM); as well as PCOS independently of the obesity factor. More scientific-based studies are required to assess whether Assisted Reproductive Technology (ART) is another predisposing factor to GDM compared to normal pregnancy.

وتعد دولة الإمارات العربية المتحدة من بين الدول العشرة الأولى في العالم من حيث السمنة ولديها أعلى معدلات متلازمة تكيس المبايض حيث تبلغ نسبتها 60% من النساء الخليجيات و30% من النساء الهنديات اللواتي يعشن في دولة الإمارات العربية المتحدة. وقد زادت السمنة جنبا إلى جنب مع زيادة تشوهات ذات الصلة في الجهاز التناسلي، مثل الإباضة والعقم. في الواقع، 1 من كل 5 أزواج في جميع أنحاء العالم يعانون من العقم، وهذا يتوافق مع 50% من النساء في دولة الإمارات العربية المتحدة حيث تواجه قضايا تتعلق العقم. تعتبر السمنة عامل خطر رئيسي لتطوير مرض السكري الحملي وكذلك تكيس المبايض وبشكل مستقل عن عامل السمنة. المزيد من الدراسات العلمية مطلوبة لتقييم ما إذا كانت التكنولوجيا المساعدة على الإنجاب عامل مؤهب آخر لمرض السكري الحملي بالمقارنة مع الحمل الطبيعي.

## Study Details

تفاصيل الدراسة

As part of this study, the researchers will measure your:

كجزء من هذه الدر اسة، فإن الباحثين سيقومون بقياس

Height

الطول ا

Weight

• الوزن

Blood pressure

و ضغط الدم

A blood sample will be collected from you at 4 episodes during your IVF treatment, which will be sent to a laboratory for the following tests:

سيتم اخذ عينة من دمك في 4 حلقات أثناء العلاج، وسيتم إرسالها إلى المختبر الإجراء الفحوصات المختبرية التالية:

• Oral Glucose Tolerance Test (OGTT)

• اختبار تحمل الجلوكوز

• Insulin level

• مستوى الأنسولين في الدم

• Women hormonal levels الشهرية الشهرية • تحليل هرمونات النساء للدورة الشهرية

• Lipid profile

• معدل الدهون

Neither the patients nor their medical insurances will be paying for these tests; but instead the ethic will be covering the costs of the tests.

It will take around two hours to complete the tests at the IVF Clinic in Dubai. There are no known risks to participate in the study and you may not benefit directly from taking part in this study. However, this study will help us assess if IVF drugs impair metabolic parameters such as glucose tolerance, insulin sensitivity and lipid profile. The study will also help screening and managing patients who are more at risk of pregnancy-related complications.

• وسوف يستغرق ساعتين لإكمال الاختبارات في مركز للإخصاب في دبي لا توجد مخاطر معروفة وقد لا تستغيد بشكل مباشر من المشاركة في هذه الدراسة . ومع ذلك، فقد تساعدنا هذه الدراسة على توضيح ما إذا كانت أدوية الإخصاب لها تأثير على المؤشرات الأيضية توازن الجلوكوز ومقاومة الانسولين ومعدل الدهون وستساعد الدراسة أيضا في فحص و رعاية المرضى الذين هم أكثر عرضة للمضاعفات المرتبطة بالحمل

All the study information will be kept confidential. You will not be identified in any publication or presentation of the study findings. Only groups' results will be reported. Blood samples (with your identification patient label code) will be preserved and stored, and can be used in the future to test other parameters. Samples will also be locked and only accessible by the PI and co-investigators. All documents from this study will be kept confidential at the IVF Clinic, locked with the principal investigator, and only accessible by the co-investigators of the study.

 و ستبقى جميع معلومات هذه الدر اسة سرية و إن يتم التعرف عليكم في أي منشور أو عرض لنتائج هذه الدر اسة سبتم حفظ وتخزين عينات الدم (مع رمز الخاص بك)، ويمكن استخدامها في المستقبل لاختبار معلمات أخرى. كما يمكن مطالعتها من قبل الباحثون في الدر اسة فقط

وسيتم إبلاغ النتائج كمجموعات فقط وسيتم الاحتفاظ بجميع الوثائق بشكل سري في مركز ويمكن مطالعتها من قبل الباحثون في الدر اسة فقط Your decision whether or not to participate will not affect your current or future relationship with the investigator, nor your IVF treatment. If you decide to participate you are free to withdraw at any time without affecting this relationship. The researchers also may choose to withdraw you from this study if this is in your interest.

• إن قرار المشاركة أو عدمه سوف لن يؤثر على علاقتك الحالية أو المستقبلية مع الباحث أو على علاجك في المركز. إذا قررت المشاركة فأنت حر في الانسحاب في أي وقت دون التأثير على هذه العلاقة وقد يكون الخيار للباحث بانسحابكم من هذه الدراسة إذا كان ذلك من مصلحتكم.

You are encouraged to ask any questions regarding this project and if you wish to find out the results of this study you may contact (contact details above) at the IVF Clinics, six months from today.

If for any ethical concern arises, you may contact the Dubai Scientific Research Ethics Committee directly (042191961/65) or by email (<u>DSREC@dha.gov.ae</u>).

• أنت مدعو لطرح أي سؤال حول هذا المشروع، وإذا كنت ترغب في معرفة نتائج هذه الدراسة عليك الاتصال (تفصيل الاتصال مذكورة أعلاه) في مركز للإخصاب وعلاج أطفال الانابيب بعد ستة أشهر من هذا البحث .

في حال نشوء أي مخاوف أخلاقية، يمكنك التواصل مع لجنة أخلاقيات البحث العلمي في دبي مباشرة ( 04219161/65) أو عن طريق البريد الإلكتروني (DSREC@dha.gov.ae

| Signed Agreement: | توقيع الاتفاق: |
|---|---|
| I understand that; | أنا أتفهم بان؛ |
| a. My signature indicates that I voluntarily agree to be a part of this | <ul> <li>أ . توقيعي يشير إلى أني أو افق طو عا على أن أكون</li> <li>جزءا من هذه الدر اسة البحثية</li> </ul> |
| research study | ب وسوف احصل على نسخة من هذا النموذج |
| b. I will receive a copy of this form | |
| Signature of Subject: | توقعٌ المشارك: |
| Date: | التاريخ: |
| Signature of Investigator: | تو قيع الباحث: |
| Date: | التاريخ: |